CLINICAL TRIAL: NCT02198781
Title: Does a Measure Exist in the Right Ventricle Which Can Act as a Surrogate Marker for Future Ventriclar Sysfunction When Pacing - a Pilot Study
Brief Title: Right Ventricle (RV) Markers of Future Pacing Induced Ventricular Dysfunction - Pilot
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: B729
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Sick Sinus Syndrome
Keywords: atrial fibrilation; atrial-ventricula; right ventricle; left ventricle; surrogate marker; ventricular dysfunction; pacing
MeSH Terms: conditions — Sick Sinus Syndrome; Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Basic science study

SUMMARY:
This is a pilot study into the effects on heart function when pacing the right ventricle (RV). This study aims to enrol a population who are clinically indicated to receive a pacemaker.

When normal conduction within the heart fails, the treatment may be to implant a permanent pacemaker. Pacing involves passing a lead via a vein to the heart and using an electrical impulse to stimulate a beat.

Increasingly the available evidence suggests that long term RV pacing is associated with complications - left ventricule (LV) dysfunction, heart failure, atrial fibrillation (AF) and death in some patients. What we do not see are a large proportion of all patients who receive pacemakers suffering pacing related adverse effects.

If there could be a way of identifying those patients in the group who go on to develop pacing induced cardiomyopathy at the time of initial pacing implant, this would be a very valuable clinical measure. These patients could be identified from the outset and paced with a biventricular device to avoid the pacing induced cardiomyopathy. Whilst much energy has been directed towards the LV as a focus of the clinical markers of disease, little has been published looking at RV haemodynamics.

We plan to study a cohort of patients who are clinically indicated to receive a pacemaker and study their RV in detail at the time of implantation. We will use conductance catheters and echocardiography to determine measures of pumping function. We will then follow them up for a period of six month using echocardiography and blood markers of heart dysfunction. In those patients who have a reduction in heart function we will then look for common patterns within their initial measurements.

DETAILED DESCRIPTION:
This study is designed to explore whether a marker exists within the right ventricle (RV) that may suggest future pacing induced dysfunction of the heart. Pacing the heart is a necessary procedure when normal conduction has failed. It has been shown in some patients to result in deleterious effects on the pumping function of the left ventricle acutely and chronically. Little has been looked into within right ventricular function and how this interacts with the left side. The fact that this dysfunction is not seen in all patients who receive pacemakers is important and we aim to use these pure haemodynamic measures to investigate this issue and try to identify those patients who may go on to have pacing induced dysfunction. This is an important scientific question to answer as we know that these patients can be spared the ventricular dysfunction by the intervention of biventricular pacing at the time of initial implantation. What we do not know is how to choose this group at the outset.

The study has been designed as a pilot investigation using patients who are to undergo permanent pacemaker therapy. Our study will entail one additional catheter being passed to the heart and also one to the inferior vena cava. This measurement of heart function will be performed directly after the implantation of the pacemaker and will add only a small amount of time to the case.

We will then follow these patients up and take echocardiographic data as well as blood markers of impaired ventricular function at 6 months.

The design of this study is that of a cohort study with the common exposure being that of pacemaker therapy. We seek to take detailed haemodynamic and echocardiographic measurements at the time of implantation. This will yield powerful data when cross referenced to cases of adverse ventricular function seen due to pacing at follow up. We aim to perform this pilot study as a feasibility process in order to ascertain the frequency of measurable adverse effects in this population and gain early insights into the markers we can look for. We do not know this data at present. This will allow for a future definitive study to be designed with appropriate participant numbers and follow up periods. The follow up period of 6 months has been set in order to fit within the time constraints of an ongoing MD undertaking.

Patients who are being booked for a pacemaker implantation as per the normal course of their treatment will be eligible to enter the study as long as they have a high anticipated pacing component. This means that these patients would be expected to have their heart stimulated via the pacemaker most of the time under normal circumstances of their care.

Patients are not eligible if they have atrial fibrillation (AF). This decision was made as patients with AF have a very different activation pattern of the heart due to the irregularity of heart rhythm and thus this would be a confounding factor to the study.

We will approach patients who meet eligibility criteria who are on the waiting list for pacemaker implantation. We will explain that this is an adjunctive procedure to the Pacemaker implant and purely for research purposes with no therapeutic benefit at the time of the procedure. We will explain the follow up needs of the study and that there potentially is a benefit to them to be followed up closely as per research protocol although this is not normal clinical workflow. Any questions will be answered at that time and consent will at a later time in preassessment clinic.

Written consent will be obtained prior to the study. The patients have the right to withdraw from the trial at any point. Consent will be verbally reconfirmed before the procedure. This process will be recorded within the medical notes at each stage.

The additional risk to the patient is insertion of the venous sheaths into the femoral vein. This is performed routinely with every electrophysiology study which is a commonly performed cardiac investigation. Very rarely the veins require to be repaired by a surgeon (1 in 500). Bleeding or bruising may occur around the sheath. Insertion of the conductance catheter into the heart may rarely (<1 in 1000) cause structural damage.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing permanent pacemaker (PPM) implantation
* Age 18-80 years old
* High grade atrial-ventricular (AV) block
* Preserved left ventricle (LV) systolic function on pre-procedure Echocardiogram (EF>45%)

Exclusion Criteria:

* Atrial Fibrillation
* Recent myocardial infarct (MI)
* Pregnancy
* Enrolment in any other study
* Inability or refusal to comply with the follow-up schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are due to undergo permanent pacemaker (PPM) implantation will be recruited to undergo RV Pressure/Volume loop assessment and RV strain ECHO at the same time as PPM implant for pilot data regarding the acute effects of RV pacing on RV haemodynamics
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
surrogate marker | 30 minutes
  To identify any surrogate markers for this patient cohort

SECONDARY OUTCOMES:
dyssynchronous index | 30 minutes
  To identify if any dyssynchronour index can be obtained in the right ventricle in this cohort

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Tan, MB BC, MRCP, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided